CLINICAL TRIAL: NCT03826719
Title: A Randomized, Double-blinded, Controlled, Phase I/II Clinical Trial to Assess the Safety, Tolerability and Immunogenicity of NBP607QIV Compared to Trivalent Egg-based Influenza Vaccine in Healty Adult Volunteers
Brief Title: Safety, Tolerability and Immunogenicity of NBP607QIV in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP607QIV_Flu_I_2013
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP607QIV (Experimental): 1 dose of 0.5mL by Intramuscular injection
  Interventions: Biological: NBP607QIV
- Agrippal (Active Comparator): 1 dose of 0.5mL by Intramuscular injection
  Interventions: Biological: Agrippal

INTERVENTIONS:
Biological: NBP607QIV — Purified inactivated influenza virus surface antigens of four strains(quadrivalent)
  Arms: NBP607QIV
Biological: Agrippal — Influenza virus surface antigens of three strains(trivalent)
  Arms: Agrippal

SUMMARY:
This study assesses safety, tolerability and immunogenicity of NBP607QIV to Agrippal which are indicated for active immunization for the prevention of influenza disease.

DETAILED DESCRIPTION:
Subjects are randomly assigned in a 1:1 ratio to NBP607QIV versus Agrippal S1. To assess the safety, solicited adverse events for 7 days post-vaccination and unsolicited adverse events for 28 days post-vaccination are assessed and reported. To assess the immunogenicity, antibody levels are evaluated by hemagglutination inhibition(HI) assay from sera obtained at pre-vaccination and 21 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 59 years
2. Those who are able and willing to give written informed consent to study participation and compliance with study instructions after being informed of and understand details of the study
3. If female, at least 2 years after post- menopausal and negative result of urine-human chorionic gonadotropin (HCG) test at screening

Exclusion Criteria:

1. Those with hypersensitivity to any component of the study medication or chemically related substances, such as allergy to eggs or egg products
2. Those with Immunodeficiency disease
3. Those with history of hypersensitivity when vaccination, such as Guillain-Barre syndrome
4. Those who are contraindicated for intramuscular injection due to thrombocytopenia or coagulopathy
5. Those who experienced fever (>38°C) within the past 24 hours or any acute respiratory infection
6. Those with history of treatment with any of Immunosuppressants or Immunomodulators within the past 3 months
7. Those with history of receiving blood products or immunoglobulin within the past 3 months
8. Those with history of influenza vaccination within the past 6 months
9. Those who received another vaccine within the past 1 month or have plan to receive another vaccine within 1 months following the study vaccination
10. Those with history of participation on another clinical trial within 1 month prior to the study vaccination
11. Those with history of blood donation within 1 week prior to the study vaccination or plan of blood donation within 7 days following the study vaccination
12. Those with any chronic diseases that interfere with the clinical trial or malignant tumors
13. Pregnant or breastfeeding
14. Those with any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or might interfere with the safety of the study subject.

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2014-03-28 (Actual); Study Completion 2014-03-28 (Actual)

PRIMARY OUTCOMES:
Incidence rate of solicited local adverse events(AEs) | 7 days after vaccination
  All AEs were classified and analyzed according to its severity and causality. The number and percentage of subjects with AEs were analyzed. Incidence rate, 95% confidence interval as well as number of occurrences were calculated.
  Comparisons within each group between pre-/post- vaccination were summarized and presented.
  The number and percentage of subjects with AEs were analyzed. Incidence rate, 95% confidence interval as well as number of occurrences were calculated.
Incidence rate of solicited systemic AEs | 7 days after vaccination
  The number and percentage of subjects with AEs were analyzed. Incidence rate, 95% confidence interval as well as number of occurrences were calculated.
Incidence rate of unsolicited AEs | 21 days after vaccination
  The number and percentage of subjects with AEs were analyzed. Incidence rate, 95% confidence interval as well as number of occurrences were calculated.

SECONDARY OUTCOMES:
Seroprotection rate measured by post-vaccination Haemagglutination Inhibition(HI) titer[Immunogenicity] | 21-28 days after vaccination
  The proportion of subjects with post-vaccination HI titers of ≥1:40
Seroconversion rate measured by pre-/post-vaccination HI titerImmunogenicity] | 21-28 days after vaccination
  The proportion of subjects achieving one of the following conditions; i)If the pre-vaccination HI titer were <1:10, subjects achieving an HI titer ≥1:40 after vaccination ii)If the pre-vaccination HI titers were ≥1:10, subjects with a minimum 4-fold rise in HI titer
9. Geometric Mean Ratio (GMR) measured by pre-/post-vaccination HI titer[Immunogenicity] | 21-28 days after vaccination
  The mean increase in geometric mean HI titer

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo Kim, MD, PhD, Study Chair — Korea University Guro Hospital

IPD SHARING:
Plan to Share IPD: No